CLINICAL TRIAL: NCT01042652
Title: A Pilot Study With Randomized Controlled Open-label Design to Compare Drug-drug Interaction, Antiretroviral Efficacy and Tolerability of Raltegravir Versus Nevirapine as Anchor Drug in Combination Therapy for Treatment-naive HIV+ Chinese Injection Drug Users on Methadone Maintenance
Brief Title: A Trial to Compare Raltegravir Versus Nevirapine as Anchor Drug for HIV+ Chinese IDUs on Methadone Maintenance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Fujie Zhang/Director, Division of Treatment and Care, NCAIDS, China CDC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X091221164
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: HIV; HIV Infections
Keywords: Methadone; HIV; Raltegravir; Antiretroviral; Intravenous Drug User; Methadone Maintenance; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nevirapine (Active Comparator)
  Interventions: Drug: Raltegravir
- Raltegravir (Experimental)
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegarvir 400mg bid

SUMMARY:
This is a pilot randomized controlled Open-label trial to compare raltegravir and nevirapine as anchor Drug in combined antiretroviral therapy(ART) for ART-naive HIV+ Chinese injection drug users who are also on methadone maintenance therapy. The investigators hypotheses include:

1. In raltegravir arm compared with nevirapine arm, fewer patients will require methadone dose adjustment to abate methadone withdrawal symptoms. Also the average methadone dose to achieve adequate serum methadone concentrations in patients on the raltegravir-based regimen will be lower compared to that of patients on the nevirapine-based regimen.
2. Clinical outcomes in terms of viral suppression, CD4 recovery and occurrence of opportunistic infections will be comparable in the two arms at 6 months and one year.
3. Patients in the raltegravir arm will have a similar or better side effect profile, retention rate, and treatment adherence compared to those in the nevirapine arm.

ELIGIBILITY:
Inclusion Criteria:

* Chinese IDUs with documented HIV-1 infection confirmed by a western blot assay.
* On stable methadone maintenance therapy at the time of enrollment.
* Antiretrovial treatment naïve and meeting clinical criteria of the Chinese national guideline to initiate antiretroviral therapy.
* Patient who is of reproductive potential agrees to use an acceptable method of birth control throughout the study. Acceptable method of birth control is defined as intrauterine device (IUD), diaphragm with spermicide, condoms, or abstinence.

Exclusion Criteria:

* Patients with allergies to or other contraindications for the selected ARV regimens.
* Patients with acute HIV infection.
* Use of concomitant therapy which can potentially interact with methadone and scheduled ARVs.
* Females who are pregnant, breast-feeding, or planning to get pregnant within the study period and using ineffective or hormonal birth control. (Note: All female patients must have a negative pregnancy test at Treatment Day 1)
* Any active and clinically significant disease or findings discovered on screening medical history, physical examination and laboratory assessment that are not resolved or stabilized within 30 days before the screening phase of this study.
* Patients with clinical or laboratory evidence of active liver disease, severe hepatic impairment /dysfunction or cirrhosis or elevated liver enzyme levels. (Note: patients co-infected with chronic hepatitis B or C will be allowed to enter the program if their condition is judged to be clinically stable.)
* Patient's education level that would interfere with the medical, adherence and withdrawal symptoms evaluation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-01 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
The percentages of patients in both arms who require methadone dose adjustment；The average methadone dose in each arm | 1 year

SECONDARY OUTCOMES:
Changes in CD4+ T lymphocyte count and viral load at weeks 24 and 48 from baseline, and the documented opportunistic infections during study period. | 1.5 year
The occurrence of side effects, adherence and retention rates in two treatment arms. | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Fujie Zhang, MD, MPH, Principal Investigator — NCAIDS, China CDC
Locations (1):
- Division of Treatment and Care, NCAIDS, China CDC, Beijing, Beijing Municipality, China